CLINICAL TRIAL: NCT06709638
Title: Clinical Evidence Based and TCM Phenotype Group Study of Zhilong Huoxue Tongyu Capsule in the Treatment of Stable Angina Pectoris of Coronary Heart Disease (Qi Deficiency and Blood Stasis Syndrome)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Jiang Hanmei (Other)
Responsible Party: Sponsor-Investigator, Jiang Hanmei, Grade 2023 master candidate of Southwest Medical University, Southwest Medical University
Organization: Southwest Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Clinical evidence based
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-02

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zhilong Huoxue Tongyu capsule (Experimental)
  Interventions: Drug: Zhilong Huoxue Tongyu capsule
- Placebo Comparator (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Other: Placebo Comparator — Placebo Comparator
  Arms: Placebo Comparator
Drug: Zhilong Huoxue Tongyu capsule — Zhilong Huoxue Tongyu capsule
  Arms: Zhilong Huoxue Tongyu capsule

SUMMARY:
This study intends to prove the clinical effect of Zhidong Huoxue Tongyu capsule in the treatment of stable angina pectoris with qi deficiency and blood stasis syndrome from the perspective of TCM syndrome differentiation and treatment. To detect metabolites in serum, urine and feces of patients with stable angina pectoris syndrome of qi deficiency and blood stasis by LC-MS metabolomics technology. Compared with normal control group, differential metabolites were found to provide molecular basis for the diagnosis of the disease. Metabolomics technology based on LC-MS was used to analyze the metabolites in serum, urine and feces before and after the treatment of Zhulong Huoxue Tongyu capsule in stable angina pectoris with qi deficiency and blood stasis syndrome. To provide laboratory evidence for Zhilong Huoxue Tongyu capsule in the treatment of stable angina pectoris with qi deficiency and blood stasis syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control group: (1) no clinical symptoms, heart color Doppler ultrasound, CTA showed no coronary heart disease and other organic heart disease; (2) Age: over 40 years old; (3) Matched with the basic information of gender, culture and education of the treatment group and the control group; (4) Voluntarily sign informed consent.

Treatment and control groups: (1) Western medicine meets the diagnostic criteria of stable angina pectoris of coronary heart disease, and there is no change in the frequency, duration, trigger or relief mode of angina pectoris attacks in the past 60 days. There was no evidence of recent myocardial injury (normal serum cardiac markers troponin T or troponin I, and no abnormal resting electrocardiogram showing significant ST-segment elevation) and angina grade I-IV. Coronary angiography or coronary CTA within 1 year: 50%< Degree of coronary artery stenosis < 75% (including left anterior descending artery, right coronary artery, left circumflex artery, and left main artery) or 50%< Degree of coronary branch vessel stenosis < 100% lesions (except main coronary arteries, such as diagonal branches). (2) consistent with TCM syndrome of Qi deficiency and blood stasis; (3) age ≥40 years old, gender is not limited; (4) Those who voluntarily sign informed consent after communication.

Exclusion Criteria:

* Healthy people: (1) liver dysfunction, renal dysfunction; (2) Participating in other clinical investigators within the past two months; (3) pregnant women, those who plan to be pregnant or lactating women.

Patients with stable angina pectoris syndrome of qi deficiency and blood stasis: (1) Those who did not meet the inclusion criteria; (2) complicated with severe hepatic and renal dysfunction; (3) pregnant and lactating women, patients with allergic constitution and a history of mental illness; (4) Acute myocardial infarction, congenital heart disease; Valvular heart disease; Myocardial infarction within the last 2 months; Patients who already have pacemakers and coronary and other stents that are not suitable for MRI materials; Malignant tumors.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
TCM syndrome integral scale | From enrollment to 60 days after treatment
CCS angina grading | From enrollment to 60 days after treatment
The number of angina attacks | From enrollment to 60 days after treatment
Nitroglycerin usage | From enrollment to 60 days after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Traditional Chinese Medicine of Southwest Medical University, Luzhou, Sichuan, China

IPD SHARING:
Plan to Share IPD: No